CLINICAL TRIAL: NCT00924664
Title: A RANDOMIZED, MULTICENTER, LONG TERM STUDY OF THE SAFETY OF TANEZUMAB IN PATIENTS WITH CHRONIC LOW BACK PAIN
Brief Title: Long Term Safety Study of Tanezumab in Chronic Low Back Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091039; CLBP SAFETY EXTENSION OF 1012 (Other: Alias Study Number)
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-03

CONDITIONS: Low Back Pain
Keywords: low back pain monoclonal antibody nerve growth factor
MeSH Terms: conditions — Low Back Pain | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tanezumab 20 mg (Experimental)
  Interventions: Biological: Tanezumab 20 mg
- Tanezumab 10 mg (Experimental)
  Interventions: Biological: Tanezumab 10 mg

INTERVENTIONS:
Biological: Tanezumab 20 mg — Tanezumab 20 mg administered IV every 8 weeks for 3 administrations followed by SC administration every 8 weeks for 4 administrations over a period of 64 weeks
  Arms: Tanezumab 20 mg
Biological: Tanezumab 10 mg — Tanezumab 10 mg administered IV every 8 weeks for 3 administrations followed by SC administration every 8 weeks for 4 administrations over a period of 64 weeks
  Arms: Tanezumab 10 mg

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of tanezumab for chronic low back pain. Patients who were randomized and treated with study medication in a previous chronic low back pain "parent" study will be eligible to enroll in this safety extension study at the Preferred Rollover Time Point visit or at the Early Termination visit of the parent study upon discontinuation due to lack of efficacy.

DETAILED DESCRIPTION:
This study was terminated on 30 November 2010 following a US FDA clinical hold for tanezumab chronic low back pain clinical studies which halted dosing and enrollment of patients on 19 July 2010 for potential safety issues.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to completing any of the study procedures.
* Female patients must meet one of the following criteria:

  1) Female patients of non childbearing potential - Must be post menopausal, defined as women who are >=45 years old with amenorrhea for 24 consecutive months (regardless of FSH levels), or women who are amenorrheic for at least 1 year AND have a serum Follicle Stimulating Hormone (FSH) level greater than 30 IU/L at Screening for the parent double blind CLBP study; or Must be surgically sterile, defined as having had a hysterectomy and/or bilateral oophorectomy.

  2.) Female patients of child bearing potential: must not be pregnant or lactating, and must be abstinent or use adequate contraception (2 forms of birth control, one of which must be a barrier method), and must have a negative serum pregnancy test at Screening (within 30 days prior to Baseline) and a negative urine pregnancy test at Baseline prior to initial dosing
* Male patients must agree that they and their female spouses / partners will use adequate contraception (2 forms of birth control, one of which must be barrier method) or be of non childbearing potential.
* Females of child bearing potential and males must be willing to use approved methods of contraception from commencement of screening procedures until 16 weeks after the last dose of IV study medication.
* Patient must be able to comply with lifestyle guidelines, scheduled visits, treatment plan, laboratory tests, and other study procedures
* Patient has been treated in a parent tanezumab double blind CLBP study
* Patient has completed the Preferred Rollover Time Point visit of the double blind CLBP parent study or has been withdrawn for lack of efficacy. At least eight weeks but no more than 12 weeks have elapsed since the last study medication infusion in the parent study. Patients are permitted to enter the extension study up to 12 weeks after their last dose of study medication in their parent study (or 4 weeks after the End of Treatment visit)

Exclusion Criteria:

* Failed screening in a parent tanezumab double blind CLBP study
* Withdrawn from a parent tanezumab double blind CLBP study for an adverse event
* Pregnant women, lactating mothers, women suspected of being pregnant, and women who wish to become pregnant during the course of clinical study
* Use of any investigational medication within 30 days prior to Baseline (3 months for any investigational biological other than tanezumab) or plans to receive an investigational medication other than the study medication during the course of this study
* Patients who exited the parent double blind CLBP study because of lack of compliance, protocol violation (including not meeting entrance criteria), no longer willing to participate (for reasons other than lack of efficacy), or were lost to follow up in the parent double blind study
* Patients who were randomized into the parent study in violation of inclusion or exclusion criteria but who were not withdrawn from the parent study;
* Any other condition, which in the opinion of the Investigator, would put the patient at increased safety risk or otherwise make the patient unsuitable for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 849 (Actual)
Dates: Start 2009-08-20 (Actual); Primary Completion 2010-11-30 (Actual); Study Completion 2011-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (149):
- United States (149):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Pinnacle Research Group, Anniston Medical Clinic, Anniston, Alabama
  - Pinnacle Research Group, Anniston, Alabama
  - Simon Williamson Clinic, PC, Birmingham, Alabama
  - Simon-Williamson Clinic, PC, Hueytown, Alabama
  - Saadat Ansari, MD, Huntsville, Alabama
  - Alabama Orthopaedic Clinic, Mobile, Alabama
  - Horizon Research Group, Mobile, Alabama
  - Phoenix Diagnostic Imaging, Chandler, Arizona
  - Radiant Research - Phoenix Southeast, Chandler, Arizona
  - Simon Med, Mesa, Arizona
  - Pivotal Research Centers, Peoria, Arizona
  - Sun Radiology, Peoria, Arizona
  - Arizona Research Center, LLC, Phoenix, Arizona
  - Radiant Research, Scottsdale, Arizona
  - Scottsdale Medical Imaging, Scottsdale, Arizona
  - Premiere Phamaceutical Research, LLC, Tempe, Arizona
  - Clinical Research Advantage, Inc./Fiel Family and Sports Medicine, PC, Tempe, Arizona
  - Little Rock Family Practice Clinic, Little Rock, Arkansas
  - Providence Clinical Research, Burbank, California
  - Valley Research, Fresno, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - University of California San Diego, La Jolla, California
  - Samaritan Center for Medical Research Medical Group, Los Gatos, California
  - Newport Diagnostic Center, Newport Beach, California
  - North County Clinical Research (NCCR), Oceanside, California
  - Advances in Medicine, Rancho Mirage, California
  - Trinity Medical Research, Roseville, California
  - Center for Clinical Trials of Sacramento, Inc., Sacramento, California
  - Wetlin Research Associates, Inc, San Diego, California
  - Inland Rheumatology & Osteoporosis Medical Group, Inc., Upland, California
  - Elite Clinical Trials, Inc., Wildomar, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Clinicos, LLC, Colorado Springs, Colorado
  - Advanced Radiology, Stamford, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - New England Research Associates, LLC, Trumbull, Connecticut
  - Southeast Clinical Research, LLC, Chiefland, Florida
  - Southeast Clinical Research, Chiefland, Florida
  - Doctors Medical Center, DeFuniak Springs, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - SJS Clinical Research, Inc., Destin, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Southeast Clinical Research, LLC, Jacksonville, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - Compass Research, LLC, Orlando, Florida
  - Palm Beach Gardens Open Imaging Center, Palm Beach Gardens, Florida
  - University Clinical Research, Pembroke Pines, Florida
  - Advent Clinical Research Center, Pinellas Park, Florida
  - Miami Research Associates, South Miami, Florida
  - Meridien Research, St. Petersburg, Florida
  - St Petersburg General Hospital - X-Rays only, St. Petersburg, Florida
  - Dale G. Bramlet, MD., P.L., St. Petersburg, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - MD Now Urgent Care, West Palm Beach, Florida
  - Midtown Imaging, West Palm Beach, Florida
  - Center for Prospective Outcome Studies, Atlanta, Georgia
  - Southeastern Radiology Associates, LLC, Atlanta, Georgia
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - CT: Marietta Imaging Center LLC, Marietta, Georgia
  - Drug Studies America, Marietta, Georgia
  - Selah Medical Center, PA, Boise, Idaho
  - Advanced Diagnostic Imaging (ADI), Evansville, Indiana
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Diagnostic Imaging Centers, Overland Park, Kansas
  - Clinical Trials Technology, Inc., Prairie Village, Kansas
  - Cotton-O'Neil Clinical Research Center, Topeka, Kansas
  - Cotton-O'Neil Clinic, Topeka, Kansas
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Commonwealth Biomedical Research, Madisonville, Kentucky
  - Arthritis and Diabetes Clinic, Monroe, Louisiana
  - Office of Peter A. Holt, MD, Baltimore, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - The Center for Clinical Trials, Biloxi, Mississippi
  - Clinical Research Center of Jackson, Jackson, Mississippi
  - Physician's Surgery Center, Jackson, Mississippi
  - Clinvest, A Division of Banyan Group, Inc, Springfield, Missouri
  - Medex Healthcare Research, Inc., St Louis, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Clinical Research Consortium, Las Vegas, Nevada
  - Mirkil Medical, Las Vegas, Nevada
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Booth Radiology, Stratford, New Jersey
  - CRI Worldwide, LLC, Willingboro, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Central New York Clinical Research, Manlius, New York
  - Medex Healthcare Research, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - B & I Imaging, Rochester, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - Greensboro Imaging, Greensboro, North Carolina
  - Pharmquest, Greensboro, North Carolina
  - Caldwell Memorial Hospital, Lenoir, North Carolina
  - Northstate Clinical Research, PLLC, Lenoir, North Carolina
  - Wake Internal Medicine Consultants, Inc., Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Christine Codding, MD, Oklahoma City, Oklahoma
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - McBride Clinic, Inc, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Medford Medical Clinic, LLP, Medford, Oregon
  - Rogue Valley Medical Center, Medford, Oregon
  - Sunstone Research, Medford, Oregon
  - Summit Research Network (Oregon), Inc., Portland, Oregon
  - Allegheny Pain Management, Altoona, Pennsylvania
  - Blair Medical Associates-Radiology, Altoona, Pennsylvania
  - Paramount Clinical Research, Bridgeville, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - CRI Worldwide LLC, Philadelphia, Pennsylvania
  - New England Center for Clinical Research, Cranston, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Columbia Arthritis Center, P.A., Columbia, South Carolina
  - Southern Orthopaedic Sports Medicine, Columbia, South Carolina
  - Radiant Research, Greer, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - SCRI Research Center, LLC, Germantown, Tennessee
  - Wolf River Medical Group, LLC, Germantown, Tennessee
  - Advanced Therapeutics, Inc., Johnson City, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - DiscoveResearch, Inc., Beaumont, Texas
  - Beaumont Internal Medicine & Geriatric Associates, Beaumont, Texas
  - DiscoveResearch Incorporated, Bryan, Texas
  - Punzi Medical Center, Carrollton, Texas
  - KRK Medical Research, Dallas, Texas
  - Advances In Health, Inc., Houston, Texas
  - St. Luke's Diagnostic & Treatment Center Kirby Glen, Houston, Texas
  - Centex Research Inc., Houston, Texas
  - Centex Research, Houston, Texas
  - Centex Research, Nassau Bay, Texas
  - Paragon Research Center, San Antonio, Texas
  - Office of Theresia Lee, MD, San Antonio, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Sendero Imaging and Treatment Center, San Antonio, Texas
  - J. Lewis Research, Inc., Salt Lake City, Utah
  - J. Lewis Research, Incorporated/Foothill Family Clinic South, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Chesapeake Regional Imaging Center-Kempsville, Norfolk, Virginia
  - Hampton Road Center for Clinical Research, Norfolk, Virginia
  - National Clinical Research - Richmond, Richmond, Virginia
  - Virginia Beach Radiology, Virginia Beach, Virginia
  - Advanced Pain Management, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Hochberg MC, Tive LA, Abramson SB, Vignon E, Verburg KM, West CR, Smith MD, Hungerford DS. When Is Osteonecrosis Not Osteonecrosis?: Adjudication of Reported Serious Adverse Joint Events in the Tanezumab Clinical Development Program. Arthritis Rheumatol. 2016 Feb;68(2):382-91. doi: 10.1002/art.39492. PMID 26554876
- [Derived] Gimbel JS, Kivitz AJ, Bramson C, Nemeth MA, Keller DS, Brown MT, West CR, Verburg KM. Long-term safety and effectiveness of tanezumab as treatment for chronic low back pain. Pain. 2014 Sep;155(9):1793-1801. doi: 10.1016/j.pain.2014.06.004. Epub 2014 Jun 14. PMID 24937440
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091039&StudyName=Long%20Term%20Safety%20Study%20of%20Tanezumab%20in%20Chronic%20Low%20Back%20Pain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who received study drug in parent study A4091012 (NCT00876187) were eligible to be enrolled in this study, either at preferred rollover visit(Day 113) or due to early discontinuation in parent study for lack of efficacy. Dosing interval between last dose in parent study and first dose in this study was not less than 8 weeks and not more than 12 weeks.
Groups:
- Tanezumab 10 mg: Participants who had previously received either tanezumab (RN624 or PF-04383119) 5, 10 milligram (mg) intravenous (IV) infusion every 8 weeks along with placebo matched to naproxen 500 mg tablet orally twice daily; or placebo matched to tanezumab IV infusion every 8 weeks along with either naproxen 500 mg tablet or matching placebo orally twice daily in parent study A4091012 (NCT00876187), received a maximum of 3 tanezumab 10 mg IV infusions over 5 minutes at 8-week interval, followed by a maximum of 3 tanezumab 10 mg subcutaneous (SC) injections at 8-week interval.
- Tanezumab 20 mg: Participants who had previously received either tanezumab (RN624 or PF-04383119) 5, 20 mg IV infusion every 8 weeks along with placebo matched to naproxen 500 mg tablet orally twice daily; or placebo matched to tanezumab IV infusion every 8 weeks along with either naproxen 500 mg tablet or matching placebo orally twice daily in parent study A4091012 (NCT00876187), received a maximum of 5 tanezumab 20 mg IV infusions over 5 minutes at 8-week interval, followed by a maximum of 3 tanezumab 20 mg SC injections at 8-week interval.
Period: Overall Study
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Started | 322 | 527
Treated | 321 | 527
Completed | 0 | 0
Not Completed | 322 | 527
Not completed — Adverse Event | 23 | 39
Not completed — Lack of Efficacy | 10 | 15
Not completed — Lost to Follow-up | 10 | 12
Not completed — Withdrawal by Subject | 47 | 71
Not completed — Protocol Violation | 2 | 5
Not completed — Pregnancy | 1 | 1
Not completed — Death | 0 | 2
Not completed — Study terminated by sponsor | 199 | 330
Not completed — Other | 29 | 52
Not completed — Randomized but not Treated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg | Total
Number analyzed (Participants) | 321 | 527 | 848
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 79 | 128 | 207
  45 to 64 years | 182 | 300 | 482
  Greater than (>) 64 years | 60 | 99 | 159
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 277 | 444
  Male | 154 | 250 | 404

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence in participant who received study medication without regard to possibility of causal relationship. SAE: AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study medication and up to 112 days after last dose that were absent before treatment in this study or that worsened relative to pretreatment state.
Time Frame: Baseline up to 112 days after last dose of study treatment (up to 448 days)
Population: Intent-to-treat (ITT) analysis set included all participants who received at least 1 dose of IV or SC study medication during this study, A4091039 (NCT00924664).
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 321 | 527
Participants
  AEs | 198 | 370
  SAEs | 15 | 24

2. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Neuropathy Impairment Score (NIS) at Week 4
Description: NIS: 74 items, assess muscle weakness, reflexes and sensation; scored separately for left, right limbs (37 items for each side). Components of muscle weakness (hip and knee flexion, hip and knee extension, ankle dorsiflexors, ankle plantar flexors, toe extensors, toe flexors) scored on scale 0 (normal) to 4 (paralysis), higher score=greater weakness. Components of reflexes (quadriceps femoris, triceps surae) and sensation (touch pressure, pin-prick, vibration, joint position) scored 0 = normal, 1= decreased, or 2 = absent. Total possible NIS score range 0-244, higher score=greater impairment.
Time Frame: A4091012: Baseline, A4091039: Week 4
Population: ITT analysis set included all participants who received at least 1 dose of IV or SC study medication during this study, A4091039 (NCT00924664). 'Number Analyzed' signifies participants evaluated at specific time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 321 | 527
units on a scale
  Baseline | 0.89 (2.53) | 1.14 (2.81)
  Change at Week 4: number analyzed (Participants) | 310 | 505
  Change at Week 4 | 0.34 (1.37) | 0.54 (2.12)

3. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Neuropathy Impairment Score (NIS) at Week 8
Description: as for outcome 2
Time Frame: A4091012: Baseline, A4091039: Week 8
Population: ITT analysis set included all participants who received at least 1 dose of IV or SC study medication during this study, A4091039 (NCT00924664). 'Overall number of participants analyzed' signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 295 | 480
units on a scale | 0.42 (1.72) | 0.54 (1.84)

4. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Neuropathy Impairment Score (NIS) at Week 16
Description: as for outcome 2
Time Frame: A4091012: Baseline, A4091039: Week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 270 | 425
units on a scale | 0.39 (1.60) | 0.42 (1.75)

5. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Neuropathy Impairment Score (NIS) at Week 24
Description: as for outcome 2
Time Frame: A4091012: Baseline, A4091039: Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 226 | 369
units on a scale | 0.35 (1.65) | 0.46 (1.93)

6. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Neuropathy Impairment Score (NIS) at Week 32
Description: as for outcome 2
Time Frame: A4091012: Baseline, A4091039: Week 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 149 | 241
units on a scale | 0.36 (1.54) | 0.32 (1.47)

7. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Neuropathy Impairment Score (NIS) at Week 40
Description: as for outcome 2
Time Frame: A4091012: Baseline, A4091039: Week 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 69 | 143
units on a scale | 0.55 (1.69) | 0.26 (1.52)

8. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Neuropathy Impairment Score (NIS) at Week 48
Description: as for outcome 2
Time Frame: A4091012: Baseline, A4091039: Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 8 | 51
units on a scale | 0.75 (2.19) | 0.18 (1.20)

9. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Neuropathy Impairment Score (NIS) at Week 56
Description: as for outcome 2
Time Frame: A4091012: Baseline, A4091039: Week 56
Population: ITT analysis set. 'Overall number of participants analyzed' signifies those participants who were evaluable for this measure. Data was not collected for tanezumab 10 mg arm at Week 56 since none of the participants received dosing beyond Week 32 and safety assessment was only required for 16 weeks after treatment discontinuation due to clinical hold.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 0 | 10
units on a scale |  | 0.70 (2.36)

10. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Brief Pain Inventory-Short Form (BPI-sf) Pain Scores (Worst, Least, Average, Right Now) at Week 4
Description: BPI-sf: 11-item self-report questionnaire consists of 5 questions, to assess severity and impact of pain on daily functions. Question/item 1-4 (Q1-Q4) measure impact of pain (worst, least, average, right now). Question 5 (Q5) consists of 7 items which measure level of interference of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life). Each item answered on 11-point scale ranging from 0 (no pain/interference) to 10 (pain as bad as you can imagine/completely interferes).
Time Frame: A4091012: Baseline, A4091039: Week 4
Population: ITT analysis set included all participants who received at least 1 dose of IV or SC study medication during this study, A4091039 (NCT00924664). 'Number Analyzed' signifies participants evaluated at specific time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 321 | 527
units on a scale
  Baseline: Worst Pain | 7.09 (1.56) | 7.29 (1.53)
  Baseline: Least Pain | 5.02 (2.09) | 4.95 (2.02)
  Baseline: Average Pain | 6.13 (1.51) | 6.25 (1.43)
  Baseline: Pain right now | 6.22 (2.01) | 6.22 (1.93)
  Change at Week 4: Worst Pain: number analyzed (Participants) | 311 | 508
  Change at Week 4: Worst Pain | -3.68 (2.65) | -3.97 (2.81)
  Change at Week 4: Least Pain: number analyzed (Participants) | 311 | 508
  Change at Week 4: Least Pain | -2.88 (2.51) | -2.93 (2.43)
  Change at Week 4: Average Pain: number analyzed (Participants) | 311 | 508
  Change at Week 4: Average Pain | -3.22 (2.39) | -3.45 (2.38)
  Change at Week 4: Pain right now: number analyzed (Participants) | 311 | 508
  Change at Week 4: Pain right now | -3.70 (2.74) | -3.86 (2.73)

11. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Brief Pain Inventory-Short Form (BPI-sf) Pain Scores (Worst, Least, Average, Right Now) at Week 8
Description: as for outcome 10
Time Frame: A4091012: Baseline, A4091039: Week 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 291 | 479
units on a scale
  Change at Week 8: Worst Pain | -3.20 (2.67) | -3.68 (2.75)
  Change at Week 8: Least Pain | -2.65 (2.49) | -2.83 (2.44)
  Change at Week 8: Average Pain | -2.92 (2.30) | -3.36 (2.36)
  Change at Week 8: Pain right now | -3.27 (2.71) | -3.63 (2.78)

12. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Brief Pain Inventory-Short Form (BPI-sf) Pain Scores (Worst, Least, Average, Right Now) at Week 16
Description: as for outcome 10
Time Frame: A4091012: Baseline, A4091039: Week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 244 | 378
units on a scale
  Change at Week 16: Worst Pain | -3.30 (2.83) | -3.58 (2.72)
  Change at Week 16: Least Pain | -2.75 (2.42) | -2.73 (2.40)
  Change at Week 16: Average Pain | -3.00 (2.41) | -3.34 (2.38)
  Change at Week 16: Pain right now | -3.42 (2.67) | -3.68 (2.67)

13. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Brief Pain Inventory-Short Form (BPI-sf) Pain Scores (Worst, Least, Average, Right Now) at Week 24
Description: as for outcome 10
Time Frame: A4091012: Baseline, A4091039: Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 155 | 258
units on a scale
  Change at Week 24: Worst Pain | -3.45 (2.80) | -3.55 (2.74)
  Change at Week 24: Least Pain | -2.79 (2.44) | -2.63 (2.34)
  Change at Week 24: Average Pain | -3.14 (2.40) | -3.31 (2.29)
  Change at Week 24: Pain right now | -3.50 (2.80) | -3.59 (2.66)

14. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Brief Pain Inventory-Short Form (BPI-sf) Pain Scores (Worst, Least, Average, Right Now) at Week 32
Description: as for outcome 10
Time Frame: A4091012: Baseline, A4091039: Week 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 68 | 128
units on a scale
  Change at Week 32: Worst Pain | -3.26 (2.90) | -3.80 (2.61)
  Change at Week 32: Least Pain | -2.50 (2.88) | -2.68 (2.35)
  Change at Week 32: Average Pain | -2.82 (2.63) | -3.23 (2.18)
  Change at Week 32: Pain right now | -3.35 (2.96) | -3.77 (2.43)

15. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Brief Pain Inventory-Short Form (BPI-sf) Pain Scores (Worst, Least, Average, Right Now) at Week 40
Description: as for outcome 10
Time Frame: A4091012: Baseline, A4091039: Week 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 8 | 37
units on a scale
  Change at Week 40: Worst Pain | -3.88 (2.42) | -3.49 (2.67)
  Change at Week 40: Least Pain | -2.75 (2.76) | -2.43 (1.91)
  Change at Week 40: Average Pain | -2.75 (3.01) | -2.97 (2.28)
  Change at Week 40: Pain right now | -3.13 (3.60) | -3.57 (2.44)

16. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Brief Pain Inventory-Short Form (BPI-sf) Pain Scores (Worst, Least, Average, Right Now) at Week 48
Description: as for outcome 10
Time Frame: A4091012: Baseline, A4091039: Week 48
Population: ITT analysis set. 'Overall number of participants analyzed' signifies those participants who were evaluable for this measure. Data was not collected for tanezumab 10 mg arm at Week 48 since none of the participants received dosing beyond Week 32 and efficacy assessment was not required after clinical hold.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 0 | 7
units on a scale
  Change at Week 48: Worst Pain |  | -2.43 (2.44)
  Change at Week 48: Least Pain |  | -0.86 (1.95)
  Change at Week 48: Average Pain |  | -2.14 (2.12)
  Change at Week 48: Pain right now |  | -2.00 (2.38)

17. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Brief Pain Inventory-Short Form (BPI-sf) Pain Scores (Worst, Least, Average, Right Now) at Week 56
Description: as for outcome 10
Time Frame: A4091012: Baseline, A4091039: Week 56
Population: Data was not collected at Week 56 since efficacy assessment was not required after clinical hold.
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 0 | 0

18. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Brief Pain Inventory-Short Form (BPI-sf) Pain Interference Scores (General Activity, Walking Ability, Normal Work, Sleep, Function Composite) at Week 4
Description: BPI-sf: 11-item self-report questionnaire consists of 5 questions, assess severity and impact of pain on daily functions. Q1-Q4 measure impact of pain (worst, least, average, right now). Q5 (7 items) measure level of interference of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). Each item answered on 11-point scale ranging from 0 (no pain/interference) to 10 (pain as bad as you can imagine/completely interferes). 7 items in Q5 averaged to obtain function composite score, range: 0 to 10; higher score=greater impairment.
Time Frame: A4091012: Baseline, A4091039: Week 4
Population: ITT analysis set included all participants who received at least 1 dose of IV or SC study medication during this study, A4091039 (NCT00924664). 'Overall number of participants analyzed' signifies those participants who were evaluable for this measure. 'Number Analyzed' signifies participants evaluated at specific time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 321 | 525
units on a scale
  Baseline: General Activity: number analyzed (Participants) | 321 | 524
  Baseline: General Activity | 5.91 (2.08) | 5.87 (2.10)
  Baseline: Walking Ability | 5.22 (2.50) | 5.40 (2.34)
  Baseline: Normal Work | 5.74 (2.18) | 5.94 (2.11)
  Baseline: Sleep | 5.97 (2.61) | 5.86 (2.50)
  Baseline: Composite score | 5.36 (2.11) | 5.37 (1.91)
  Change at Week 4: General Activity: number analyzed (Participants) | 311 | 505
  Change at Week 4: General Activity | -3.39 (2.76) | -3.45 (2.81)
  Change at Week 4: Walking Ability: number analyzed (Participants) | 311 | 506
  Change at Week 4: Walking Ability | -2.85 (2.88) | -3.15 (2.85)
  Change at Week 4: Normal Work: number analyzed (Participants) | 311 | 506
  Change at Week 4: Normal Work | -3.15 (2.71) | -3.49 (2.80)
  Change at Week 4: Sleep: number analyzed (Participants) | 311 | 506
  Change at Week 4: Sleep | -3.53 (3.13) | -3.45 (2.98)
  Change at Week 4: Composite score: number analyzed (Participants) | 311 | 506
  Change at Week 4: Composite score | -3.09 (2.52) | -3.21 (2.45)

19. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Brief Pain Inventory-Short Form (BPI-sf) Pain Interference Scores (General Activity, Walking Ability, Normal Work, Sleep, Function Composite) at Week 8
Description: as for outcome 18
Time Frame: A4091012: Baseline, A4091039: Week 8
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 291 | 478
units on a scale
  Change at Week 8: General Activity: number analyzed (Participants) | 291 | 477
  Change at Week 8: General Activity | -2.99 (2.65) | -3.36 (2.88)
  Change at Week 8: Walking Ability | -2.58 (2.68) | -3.00 (2.89)
  Change at Week 8: Normal Work: number analyzed (Participants) | 290 | 478
  Change at Week 8: Normal Work | -2.77 (2.62) | -3.32 (2.90)
  Change at Week 8: Sleep | -3.15 (3.06) | -3.34 (2.96)
  Change at Week 8: Composite score | -2.74 (2.40) | -3.09 (2.52)

20. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Brief Pain Inventory-Short Form (BPI-sf) Pain Interference Scores (General Activity, Walking Ability, Normal Work, Sleep, Function Composite) at Week 16
Description: as for outcome 18
Time Frame: A4091012: Baseline, A4091039: Week 16
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 244 | 376
units on a scale
  Change at Week 16: General Activity: number analyzed (Participants) | 244 | 375
  Change at Week 16: General Activity | -3.20 (2.81) | -3.26 (2.89)
  Change at Week 16: Walking Ability | -2.55 (2.76) | -2.94 (2.93)
  Change at Week 16: Normal Work: number analyzed (Participants) | 244 | 375
  Change at Week 16: Normal Work | -2.83 (2.61) | -3.26 (2.84)
  Change at Week 16: Sleep | -3.19 (2.93) | -3.34 (2.94)
  Change at Week 16: Composite score | -2.76 (2.44) | -3.05 (2.51)

21. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Brief Pain Inventory-Short Form (BPI-sf) Pain Interference Scores (General Activity, Walking Ability, Normal Work, Sleep, Function Composite) at Week 24
Description: as for outcome 18
Time Frame: A4091012: Baseline, A4091039: Week 24
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 155 | 256
units on a scale
  Change at Week 24: General Activity | -3.12 (2.87) | -3.25 (2.95)
  Change at Week 24: Walking Ability: number analyzed (Participants) | 154 | 256
  Change at Week 24: Walking Ability | -2.70 (2.84) | -2.90 (2.81)
  Change at Week 24: Normal Work | -3.06 (2.80) | -3.25 (2.77)
  Change at Week 24: Sleep: number analyzed (Participants) | 154 | 256
  Change at Week 24: Sleep | -3.47 (2.91) | -3.42 (2.96)
  Change at Week 24: Composite score | -2.90 (2.52) | -3.03 (2.50)

22. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Brief Pain Inventory-Short Form (BPI-sf) Pain Interference Scores (General Activity, Walking Ability, Normal Work, Sleep, Function Composite) at Week 32
Description: as for outcome 18
Time Frame: A4091012: Baseline, A4091039: Week 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 68 | 127
units on a scale
  Change at Week 32: General Activity | -2.47 (3.21) | -3.17 (2.67)
  Change at Week 32: Walking Ability | -2.32 (3.26) | -2.74 (2.78)
  Change at Week 32: Normal Work | -2.74 (3.31) | -3.20 (2.65)
  Change at Week 32: Sleep | -3.10 (3.22) | -3.47 (2.91)
  Change at Week 32: Composite score | -2.52 (3.09) | -2.94 (2.32)

23. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Brief Pain Inventory-Short Form (BPI-sf) Pain Interference Scores (General Activity, Walking Ability, Normal Work, Sleep, Function Composite) at Week 40
Description: as for outcome 18
Time Frame: A4091012: Baseline, A4091039: Week 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 8 | 37
units on a scale
  Change at Week 40: General Activity | -2.88 (3.04) | -2.46 (2.55)
  Change at Week 40: Walking Ability | -2.13 (2.53) | -2.59 (2.73)
  Change at Week 40: Normal Work | -2.63 (3.38) | -2.73 (2.36)
  Change at Week 40: Sleep | -3.13 (3.72) | -3.41 (2.62)
  Change at Week 40: Composite score | -2.27 (3.18) | -2.72 (2.28)

24. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Brief Pain Inventory-Short Form (BPI-sf) Pain Interference Scores (General Activity, Walking Ability, Normal Work, Sleep, Function Composite) at Week 48
Description: as for outcome 18
Time Frame: A4091012: Baseline, A4091039: Week 48
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 0 | 7
units on a scale
  Change at Week 48: General Activity |  | -1.71 (2.21)
  Change at Week 48: Walking Ability |  | -1.71 (2.21)
  Change at Week 48: Normal Work |  | -1.57 (1.99)
  Change at Week 48: Sleep |  | -2.43 (1.13)
  Change at Week 48: Composite score |  | -1.76 (1.53)

25. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Brief Pain Inventory-Short Form (BPI-sf) Pain Interference Scores (General Activity, Walking Ability, Normal Work, Sleep, Function Composite) at Week 56
Description: as for outcome 18
Time Frame: A4091012: Baseline, A4091039: Week 56
Population: Data was not collected at Week 56 since efficacy assessment was not required after clinical hold.
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 0 | 0

26. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Roland-Morris Disability Questionnaire (RMDQ) Total Score at Week 4
Description: RMDQ: back-specific, participant administered questionnaire that assess how well participants with low back pain were able to function with regard to daily activities. The questionnaire consists of 24 statements and the participant is instructed to put a mark next to each appropriate statement. The number of statements marked are added up by the clinician. Total RMDQ score was calculated as the sum of number of statements checked. Total possible RMDQ score: 0 to 24, with higher scores indicated greater disability.
Time Frame: A4091012: Baseline, A4091039: Week 4
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 320 | 525
units on a scale
  Baseline | 13.01 (5.13) | 12.66 (4.85)
  Change at Week 4: number analyzed (Participants) | 256 | 419
  Change at Week 4 | -5.52 (5.73) | -5.35 (5.47)

27. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Roland-Morris Disability Questionnaire (RMDQ) Total Score at Week 8
Description: RMDQ: back-specific, participant administered questionnaire that assess how well participants with low back pain were able to function with regard to daily activities. The questionnaire consists of 24 statements and the participant is instructed to put a mark next to each appropriate statement. The number of statements marked are added up by the clinician. Total RMDQ score is calculated as the sum of number of statements checked. Total possible RMDQ score: 0 to 24, with higher scores indicated greater disability.
Time Frame: A4091012: Baseline, A4091039: Week 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 245 | 399
units on a scale | -4.86 (5.14) | -5.02 (5.71)

28. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Roland-Morris Disability Questionnaire (RMDQ) Total Score at Week 16
Description: as for outcome 27
Time Frame: A4091012: Baseline, A4091039: Week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 202 | 310
units on a scale | -4.90 (5.84) | -5.19 (5.36)

29. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Roland-Morris Disability Questionnaire (RMDQ) Total Score at Week 24
Description: as for outcome 27
Time Frame: A4091012: Baseline, A4091039: Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 126 | 210
units on a scale | -4.79 (5.64) | -5.30 (5.61)

30. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Roland-Morris Disability Questionnaire (RMDQ) Total Score at Week 32
Description: as for outcome 27
Time Frame: A4091012: Baseline, A4091039: Week 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 59 | 107
units on a scale | -5.36 (5.87) | -5.07 (5.46)

31. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Roland-Morris Disability Questionnaire (RMDQ) Total Score at Week 40
Description: as for outcome 27
Time Frame: A4091012: Baseline, A4091039: Week 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 8 | 32
units on a scale | -6.00 (6.32) | -4.13 (6.32)

32. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Roland-Morris Disability Questionnaire (RMDQ) Total Score at Week 48
Description: as for outcome 27
Time Frame: A4091012: Baseline, A4091039: Week 48
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 0 | 6
units on a scale |  | -2.67 (6.02)

33. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Roland-Morris Disability Questionnaire (RMDQ) Total Score at Week 56
Description: as for outcome 27
Time Frame: A4091012: Baseline, A4091039: Week 56
Population: Data was not collected at Week 56 since efficacy assessment was not required after clinical hold.
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 0 | 0

34. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Patient Global Assessment of Low Back Pain at Week 4
Description: Participants answered: "Considering all ways your low back pain affects you, how are you doing today?" Participants rated their condition using scale assessing symptoms and limitations to carry out normal daily activities. Score range: 1-5. 1: Very Good (No symptoms and limitations); 2: Good (Mild symptoms and no limitations); 3: Fair (Moderate symptoms and some limitations); 4: Poor (Severe symptoms and inability to carry out most activities); 5: Very Poor (Very severe, intolerable symptoms and inability to carry all activities).
Time Frame: A4091012: Baseline, A4091039: Week 4
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 321 | 527
units on a scale
  Baseline | 3.38 (0.57) | 3.36 (0.56)
  Change at Week 4: number analyzed (Participants) | 310 | 508
  Change at Week 4 | -1.17 (1.00) | -1.21 (1.00)

35. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Patient Global Assessment of Low Back Pain at Week 8
Description: as for outcome 34
Time Frame: A4091012: Baseline, A4091039: Week 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 291 | 480
units on a scale | -0.97 (0.97) | -1.07 (1.01)

36. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Patient Global Assessment of Low Back Pain at Week 16
Description: as for outcome 34
Time Frame: A4091012: Baseline, A4091039: Week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 244 | 376
units on a scale | -1.05 (1.02) | -1.03 (0.96)

37. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Patient Global Assessment of Low Back Pain at Week 24
Description: as for outcome 34
Time Frame: A4091012: Baseline, A4091039: Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 154 | 258
units on a scale | -1.09 (0.95) | -1.05 (1.01)

38. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Patient Global Assessment of Low Back Pain at Week 32
Description: as for outcome 34
Time Frame: A4091012: Baseline, A4091039: Week 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 68 | 128
units on a scale | -1.07 (1.14) | -1.05 (0.98)

39. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Patient Global Assessment of Low Back Pain at Week 40
Description: as for outcome 34
Time Frame: A4091012: Baseline, A4091039: Week 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 8 | 37
units on a scale | -1.25 (1.04) | -0.95 (1.03)

40. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Patient Global Assessment of Low Back Pain at Week 48
Description: as for outcome 34
Time Frame: A4091012: Baseline, A4091039: Week 48
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 0 | 7
units on a scale |  | -0.43 (0.79)

41. Primary Outcome: Change From A4091012 (NCT00876187) Baseline in Patient Global Assessment of Low Back Pain at Week 56
Description: as for outcome 34
Time Frame: A4091012: Baseline, A4091039: Week 56
Population: Data was not collected at Week 56 since efficacy assessment was not required after clinical hold.
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 0 | 0

42. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Description: Median time to discontinuation due to lack of efficacy was estimated using Kaplan-Meier method.
Time Frame: Baseline up to Week 56
Population: ITT analysis set included all participants who received at least 1 dose of IV or SC study medication during this study, A4091039 (NCT00924664).
Measure: Median (Full Range); unit: days
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 321 | 527
days | NA [NA to NA] — Median and full range were not evaluable since very few participants discontinued due to lack of efficacy. | NA [NA to NA] — Median and full range were not evaluable since very few participants discontinued due to lack of efficacy.

43. Secondary Outcome: Plasma Concentration of Tanezumab
Description: Analysis was done by setting concentration values below the lower limit of quantification (LLOQ) to zero.
Time Frame: Baseline (Day 1), Week 8, 24, 40, 56, 64
Population: Pharmacokinetic(PK) analysis set: participants who received at least 1 dose of IV or SC study medication during this study, A4091039(NCT00924664), had at least 1 plasma concentration value above LLOQ. 'Overall Number of Participants Analyzed' signifies participants evaluable for this measure, 'Number Analyzed' signifies participants evaluated at specific time points for each arm group, respectively. Due to clinical hold, study was terminated prematurely, data was not collected at Week 64.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 268 | 433
nanogram/milliliter (ng/mL)
  Baseline: number analyzed (Participants) | 62 | 96
  Baseline | 393.519 (659.8150) | 427.871 (771.2499)
  Week 8 | 596.957 (533.8274) | 1074.76 (527.5588)
  Week 24: number analyzed (Participants) | 150 | 248
  Week 24 | 588.216 (296.7509) | 1276.75 (770.0278)
  Week 40: number analyzed (Participants) | 7 | 48
  Week 40 | 542.571 (240.5285) | 1058.92 (666.4789)
  Week 56: number analyzed (Participants) | 238 | 396
  Week 56 | 250.512 (393.9501) | 502.320 (676.1049)

44. Secondary Outcome: Total Nerve Growth Factor (NGF) Concentration
Time Frame: Baseline (Day 1), Week 8, 24, 40, 56, 64
Population: ITT analysis set. 'Overall number of participants analyzed' signifies participants evaluable for this measure. 'Number Analyzed' signifies participants evaluated at specific time points for each arm group, respectively. Data was not collected at Week 64 since assessment was only required for 16 weeks after treatment discontinuation due to clinical hold.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 270 | 430
picogram/milliliter
  Baseline: number analyzed (Participants) | 57 | 76
  Baseline | 2599.9 (1893.7) | 2025.4 (2281.4)
  Week 8 | 3771.1 (1472.3) | 4470.2 (1773.6)
  Week 24: number analyzed (Participants) | 149 | 249
  Week 24 | 4132.7 (1780.1) | 4860.6 (1990.6)
  Week 40: number analyzed (Participants) | 7 | 46
  Week 40 | 4314.0 (1372.4) | 4446.7 (1807.1)
  Week 56: number analyzed (Participants) | 233 | 387
  Week 56 | 2855.5 (1651.8) | 3639.3 (1990.3)

45. Other Pre Specified Outcome: Number of Participants Using Concomitant Medication for Chronic Low Back Pain (CLBP)
Description: Food and Drug Administration (FDA) approved analgesics and muscle relaxants were permitted as concomitant medications for CLBP and were prescribed as per investigator's discretion. These medications included opioids, topical analgesics, non-steroidal anti-inflammatory drug (NSAIDs), capsaicin products, oral/injectable corticosteroids, and viscosupplementation (eg, hyaluronan).
Time Frame: Baseline up to Week 56
Population: as for outcome 42
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 321 | 527
Participants | 150 | 268

46. Other Pre Specified Outcome: Change From A4091012 (NCT00876187) Baseline in Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) at Week 24 and 56
Description: WPAI:SHP: 6-item, binary question on current employment, 3 questions on hours of work and work-loss, 2 questions based on 0-10 point scale to judge how CLBP affects ability to work, perform regular activities(0=no effect on work/activity, 10=completely prevented from working/activity). Four scores derived as percent: activity impairment, impairment while working, overall work impairment, work time missed. Total possible score: 0-100 (0=no impairment/high productivity, 100=completely impaired/low activity). Each of 4 scores expressed as impairment percentages, high percentage=more impairment, less productivity.
Time Frame: A4091012: Baseline, A4091039: Week 24, 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 321 | 527
percentage of impairment
  Baseline:activity impairment: number analyzed (Participants) | 321 | 523
  Baseline:activity impairment | 58.19 (23.05) | 58.74 (21.24)
  Baseline:impairment during work: number analyzed (Participants) | 163 | 277
  Baseline:impairment during work | 48.77 (23.56) | 47.98 (23.66)
  Baseline:overall impairment | 8.23 (23.11) | 7.46 (21.97)
  Baseline:work time missed | 2.99 (10.81) | 2.27 (8.67)
  Change at Week 24:activity impairment: number analyzed (Participants) | 204 | 344
  Change at Week 24:activity impairment | -25.29 (27.64) | -26.34 (28.55)
  Change at Week 24:impairment during work: number analyzed (Participants) | 92 | 154
  Change at Week 24:impairment during work | -26.30 (24.79) | -21.36 (26.84)
  Change at Week 24:overall impairment: number analyzed (Participants) | 221 | 364
  Change at Week 24:overall impairment | -4.63 (23.62) | -3.25 (21.39)
  Change at Week 24:work time missed: number analyzed (Participants) | 221 | 364
  Change at Week 24:work time missed | -1.49 (10.33) | -0.50 (8.24)
  Change at Week 56:activity impairment: number analyzed (Participants) | 0 | 10
  Change at Week 56:activity impairment |  | -8.00 (34.58)
  Change at Week 56:impairment during work: number analyzed (Participants) | 0 | 6
  Change at Week 56:impairment during work |  | -10.00 (28.28)
  Change at Week 56:overall impairment: number analyzed (Participants) | 0 | 10
  Change at Week 56:overall impairment |  | 1.75 (16.76)
  Change at Week 56:work time missed: number analyzed (Participants) | 0 | 10
  Change at Week 56:work time missed |  | 1.41 (4.71)

47. Other Pre Specified Outcome: Number of Participants Who Developed Anti-Tanezumab Antibodies
Description: Human serum anti-drug antibody (ADA) samples were analyzed for the presence or absence of anti-tanezumab antibodies by using the semi-quantitative enzyme-linked immunosorbent assay (ELISA). Same participant may have positive ADA result at more than 1 time point.
Time Frame: Baseline (Day 1), Week 8, 24, 40, 56, 64
Population: ITT analysis set. 'Overall number of participants analyzed'=participants evaluable for this measure at any time point. 'Number Analyzed' signifies participants evaluated at specific time points for each arm, respectively. Data was not analyzed at Week 64 since safety assessment was only required for 16 weeks after treatment discontinuation due to clinical hold.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 269 | 435
Participants
  Baseline: number analyzed (Participants) | 61 | 96
  Baseline | 1 | 0
  Week 8 | 4 | 1
  Week 24: number analyzed (Participants) | 153 | 252
  Week 24 | 3 | 1
  Week 40: number analyzed (Participants) | 7 | 48
  Week 40 | 0 | 0
  Week 56: number analyzed (Participants) | 237 | 396
  Week 56 | 1 | 1

48. Other Pre Specified Outcome: Number of Participants With Injection and Infusion Site Reactions
Description: The injection and infusion site reactions were assessed based on presence of erythema (redness), induration (swelling), ecchymosis (bruising), pruritus (itching) and pain that occurred after administration (not related to needle insertion pain) of subcutaneous injection or intravenous infusion.
Time Frame: Baseline (Day 1), Week 4, 8, 16, 24, 32 for intravenous infusion; Week 24, 32, 40, 56, 64 for subcutaneous injection
Population: ITT analysis set. Data was not analyzed at Week 64 for SC injection since safety assessment was only required for 16 weeks after treatment discontinuation due to clinical hold.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 321 | 527
Participants
  Baseline: Infusion site | 7 | 7
  Week 4: Infusion site | 0 | 0
  Week 8: Infusion site | 5 | 5
  Week 16: Infusion site | 4 | 5
  Week 24: Infusion site | 0 | 0
  Week 32: Infusion site | 0 | 0
  Week 24: Injection site | 2 | 4
  Week 32: Injection site | 0 | 2
  Week 40: Injection site | 0 | 0
  Week 56: Injection site | 0 | 0

49. Other Pre Specified Outcome: Number of Participants With Intravenous and Subcutaneous Doses of Study Medication
Description: Number of participants are reported based on the maximum number of intravenous (IV) and subcutaneous (SC) doses of tanezumab received.
Time Frame: Day 1 up to Week 56
Population: as for outcome 42
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 321 | 527
Participants
  Number of IV Doses: 1 | 59 | 102
  Number of IV Doses: 2 | 93 | 145
  Number of IV Doses: 3 | 169 | 276
  Number of IV Doses: 4 | 0 | 3
  Number of IV Doses: 5 | 0 | 1
  Number of SC Doses: 1 | 71 | 111
  Number of SC Doses: 2 | 8 | 42
  Number of SC Doses: 3 | 1 | 7

ADVERSE EVENTS:
Description: Cases of osteonecrosis (ON) reported in this and other studies conducted up to 2010 were adjudicated post-hoc by an expert committee (2010-2012). Few of these events (2 of 87 reported ON cases), were confirmed as ON by the committee. Source: https://doi.org/10.1002/art.39492
Arm/Group | Tanezumab 10 mg | Tanezumab 20 mg
Serious Adverse Events (participants affected / at risk) | 15/321 | 24/527
Other Adverse Events (participants affected / at risk) | 152/321 | 277/527
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 10 mg (N=321) | Tanezumab 20 mg (N=527)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 3
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 10 mg (N=321) | Tanezumab 20 mg (N=527)
Diarrhoea (Gastrointestinal disorders) | 6 | 18
Infusion site reaction (General disorders) | 12 | 17
Oedema peripheral (General disorders) | 11 | 32
Nasopharyngitis (Infections and infestations) | 5 | 13
Sinusitis (Infections and infestations) | 12 | 14
Upper respiratory tract infection (Infections and infestations) | 11 | 26
Urinary tract infection (Infections and infestations) | 9 | 13
Fall (Injury, poisoning and procedural complications) | 7 | 15
Muscle strain (Injury, poisoning and procedural complications) | 8 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 41 | 76
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 17
Joint swelling (Musculoskeletal and connective tissue disorders) | 6 | 16
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 15
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 | 22
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 18
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 38
Allodynia (Nervous system disorders) | 0 | 11
Decreased vibratory sense (Nervous system disorders) | 2 | 14
Headache (Nervous system disorders) | 10 | 27
Hyperaesthesia (Nervous system disorders) | 3 | 11
Hypoaesthesia (Nervous system disorders) | 23 | 41
Paraesthesia (Nervous system disorders) | 31 | 56
Rash (Skin and subcutaneous tissue disorders) | 2 | 11

LIMITATIONS AND CAVEATS:
Due to FDA-imposed clinical hold, further study drug dosing stopped prematurely and study was terminated. Designation of outcomes as primary, secondary based on study team input as study did not specify them as primary or secondary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.